CLINICAL TRIAL: NCT04671784
Title: Endoscopic Ultrasound Elastography (Strain Ratio) and Fractal-based Quantitative Analysis for the Mediastinal and Abdominal Lymphadenopathies
Acronym: Lymph/EUS/01
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2364
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Lymph Nodes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Enlarged mediastinal or abdominal: Consecutive patients with enlarged mediastinal or abdominal detected by cross-sectional imaging and confirmed at EUS will be enrolled.
  Interventions: Other: EUS-E

INTERVENTIONS:
Other: EUS-E — EUS-E

SUMMARY:
Endoscopic ultrasound (EUS) and EUS-guided tissue acquisition (EUS-TA) are minimally invasive techniques to establish the benign or malignant nature of lymph nodes (LNs) with a very high accuracy. In particular, for mediastinal LNs, a meta-analysis underlined that EUS features alone are not enough to reach a good sensitivity and specificity, while EUS-TA showed a slightly high sensitivity (88% vs. 85%) and a significantly high specificity (96% vs. 85%) for diagnosing the cause of LN enlargement. Considering all sites, according to the meta-analysis of Xu and colleagues, the assessment of LNs by EUS-elastography is a useful tool in differentiating benign and malignant LNs, with a sensitivity of 88% and a specificity of 85%.

For lymphadenopathy of unknown origin, ESGE recommends performing EUS-TA (or alternatively endobronchial ultrasound [EBUS]-guided) if the patient management requires a pathological result and no superficial lymphadenopathy is easily accessible. Unfortunately, EUS-TA may sometimes be challenging or inconclusive, due to blood contamination or insufficient material.

EUS elastography (EUS-E) is a non-invasive ultrasound technique that measures the hardness of tissues. The level of hardness of region of interest (ROI) can be evaluated using qualitative scores and/or quantitative methods (strain ratio; SR).

To date, most of the studies on EUS-E have been carried out using the Hitachi ultrasound machine. In particular, Paterson performed a quantitative analysis considering as a pathological value cut-off, the SR ≥7.5 for EUS-E in the nodal staging of esophageal cancer. The study involved 53 LNs using cytology as gold standard: their data showed that EUS-E had a sensitivity of 83%, specificity of 96%, PPV of 95% and NPV of 86%.

Recently, a new compact ultrasound processor, EU-ME2 (Olympus SE & CO. KG, Hamburg, Germany) that includes an elastography software was developed although data regarding its application in LNs evaluation are still not available. The concept of fractal geometry as a tool for describing natural objects was originally introduced by Benoit Mandelbrot. A fractal can be considered as an irregularly shaped object and that can be divided into fragments, each of them representing a self-similar reduced copy of the whole. The hun body is an example of natural fractal, as many of its parts are characterized by features resembling the typical fractal nature. It has been demonstrated that fractal geometry can be used to efficiently evaluate the geometrical complexity of imaging patterns observed in oncology.

The investigators recently published a study on the role of EUS elastography and fractal based analysis in the differentiation of solid pancreatic lesions. However, data regarding the application of fractal analysis to evaluate lymphadenopathies are still not available.

ELIGIBILITY:
Inclusion Criteria:

* patients with identified enlarged lymph nodes;
* patients >18 years old.

Exclusion Criteria:

* patients who decline to participate in the study
* patients with contraindication to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with enlarged mediastinal or abdominal lymph nodes detected by cross-sectional imaging and confirmed at EUS will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of quantitative EUS-E (strain ratio) | 24 Months
  The primary aim of this study is to evaluate the accuracy of quantitative EUS-E (strain ratio) for the diagnosis of malignancy in enlarged lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No